CLINICAL TRIAL: NCT02085499
Title: Effects of Flow-synchronized Nasal Intermittent Mandatory Ventilation in Preterm Infants
Brief Title: Flow-synchronized Nasal IMV in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Nelson Claure, Research Associate Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20130844
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Premature Infant Disease; Respiratory Insufficiency
Keywords: nasal ventilation; premature infants; synchronized ventilation; non-invasive respiratory support
MeSH Terms: conditions — Respiratory Insufficiency; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIMV followed by S-NIMV (Other): During the study infants assigned to this arm will undergo a 2-hour period of non-synchronized NIMV followed by a 2-hour period of Synchronized-NIMV.
  Interventions: Other: non-synchronized NIMV; Other: Synchronized NIMV
- S-NIMV followed by NIMV (Other): During the study infants assigned to this arm will undergo a 2-hour period of synchronized NIMV followed by a 2-hour period of non-synchronized NIMV.
  Interventions: Other: non-synchronized NIMV; Other: Synchronized NIMV

INTERVENTIONS:
Other: non-synchronized NIMV — During the study each infant will undergo a 2-hour period of NIMV at a frequency of 30 cycles per minute.
  NIMV will be provided by a time cycled, pressure limited neonatal ventilator (Puritan Bennett 840, Covidien, Boulder, CO).
Other: Synchronized NIMV — During the study each infant will undergo a 2-hour period of S-NIMV at a frequency of 30 cycles per minute.
  S-NIMV will be provided by a time cycled, pressure limited neonatal ventilator, with leak compensation capacity and nasal flow triggered ventilation (Puritan Bennett 840, Covidien, Boulder, CO). Synchronization will be achieved by the leak compensation software and the internal sensor of the ventilator.

SUMMARY:
The use of non-invasive methods of respiratory support to reduce complications of prolonged invasive mechanical ventilation in preterm infants has increased.

The most common mode is nasal intermittent mandatory ventilation (NIMV). In NIMV, the interval between mechanical breaths is fixed and is determined by the frequency dialed by the clinician. Asynchrony between the infant's spontaneous breathing may exist since mechanical breaths delivered at fixed intervals can occur at different times over the inspiratory or expiratory phases of the infant's spontaneous breathing. Synchronized-NIMV is a mode similar to NIMV where the ventilator cycle is delivered in synchrony with the infant's spontaneous inspiration. This has been achieved by using techniques to detect the infant's spontaneous inspiration.

The advantages or disadvantages of synchronized compared to non-synchronized NIMV remain to be determined.

This study seeks to evaluate the effect of synchronized NIMV versus non-synchronized NIMV on ventilation and gas exchange in premature infants who require supplemental oxygen.

The hypothesis is that the use of flow synchronized nasal intermittent mandatory ventilation (S-NIMV) in comparison to non-synchronized NIMV will improve ventilation and gas exchange and reduce breathing effort.

The objective of the study is to compare the effect of flow synchronized-NIMV to non-synchronized-NIMV on tidal volume (VT), minute ventilation (VE), gas exchange, breathing effort, apnea and chest wall distortion in preterm neonates with lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants of 30 or less weeks of gestational age
* Receiving NIMV
* Requiring Fi02 > 0.21 to keep Sp02 > 90%
* Parental written informed consent

Exclusion Criteria:

* Major congenital anomalies
* Proven sepsis within 72 hours of the study
* Hypotension requiring pressors within 72 hours of the study
* Pneumothorax or pneumomediastinum within 72 hours of the study
* Current suspected necrotizing enterocolitis, spontaneous perforation or severe abdominal distention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Minute Ventilation | 4 hours
  Measurements of minute ventilation (VE in ml-units/min/Kg) by respiratory inductance plethysmography during flow synchronized-NIMV will be compared to measurements during non-synchronized-NIMV
Ttidal volume (VT) | 4 hours
  Measurements of tidal volume (VT in ml-units/Kg) by respiratory inductance plethysmography during flow synchronized-NIMV will be compared to measurements during non-synchronized-NIMV

SECONDARY OUTCOMES:
Arterial oxygen saturation | 4 hours
  Measurements of arterial oxygen saturation (%) by pulse oximetry obtained during flow synchronized-NIMV will be compared to measurements obtained during non-synchronized-NIMV
fraction of inspired oxygen | 4 hours
  Required fraction of inspired oxygen during flow synchronized-NIMV will be compared to measurements obtained during non-synchronized-NIMV
transcutaneous carbon dioxide tension | 4 hours
  Measurements of transcutaneous carbon dioxide tension (mmHg) obtained during flow synchronized-NIMV will be compared to measurements obtained during non-synchronized-NIMV

OTHER OUTCOMES:
Inspiratory breathing effort | 4 hours
  Measurements of inspiratory breathing effort obtained by esophageal manometry (cmH2O) during flow synchronized-NIMV will be compared to measurements obtained during non-synchronized-NIMV
Chest wall distortion by Tcd/Vt ratio | 4 hours
  Measurements of inspiratory chest wall distortion (Tcd/Vt ratio) obtained during flow synchronized-NIMV will be compared to measurements obtained during non-synchronized-NIMV
Chest wall distortion by phase lag | 4 hours
  Measurements of inspiratory chest wall distortion (phase lag in degrees) obtained during flow synchronized-NIMV will be compared to measurements obtained during non-synchronized-NIMV
apnea frequency | 4 hours
  Measurements of apneic respiratory pauses (#/hour) obtained during flow synchronized-NIMV will be compared to measurements obtained during non-synchronized-NIMV

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Claure, MSc, PhD, Principal Investigator — University of Miami; Eduardo Bancalari, MD, Principal Investigator — University of Miami
Locations (1):
- Holtz Childrens Hospital-Jackson Health System-University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No